CLINICAL TRIAL: NCT03727061
Title: A Phase 1 Trial: Porfimer Sodium Mediated Interstitial Photodynamic for the Treatment of Patients With Locally Advanced or Recurrent Head and Neck Cancer
Brief Title: Porfimer Sodium Interstitial Photodynamic Therapy With or Without Standard of Care Chemotherapy in Treating Patients With Locally Advanced or Recurrent Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 67918; R01CA193610 (NIH); P01CA055791 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Head and Neck Carcinoma; Locally Advanced Head and Neck Carcinoma
MeSH Terms: interventions — Nivolumab; Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm A(porfimer sodium, I-PDT (Experimental): Patients receive porfimer sodium IV over 3-5 minutes and undergo I-PDT approximately 48 hours later.
  Interventions: Biological: Nivolumab; Drug: Porfimer Sodium; Procedure: Interstitial Illumination Photodynamic Therapy; Other: Quality of Life Assessment

INTERVENTIONS:
Biological: Nivolumab — Immunotherapy - Standard of care
  Other Names: NIVO, NIVOLUMAB, Nivolumab, BMS-936558
Drug: Porfimer Sodium — Given IV
  Other Names: Photofrin II, Photofrin II, PORFIMER SODIUM, porfimer sodium, Porfimer Sodium
Procedure: Interstitial Illumination Photodynamic Therapy — Undergo I-PDT
Other: Quality of Life Assessment — Ancillary Studies

SUMMARY:
This phase I trial studies the side effects of interstitial photodynamic therapy (I-PDT) in treating patients with head and neck cancer that has spread to other parts of the body or that has come back. Interstitial photodynamic therapy uses a light-sensitive drug called porfimer sodium. This drug is activated by laser light delivered through special fibers into the tumor.

In this study the doctors will evaluate the safety of I-PDT and determine the potentially effective light setting in this treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of porfimer sodium (Photofrin) mediated interstitial photodynamic therapy (I-PDT) in patients with locally advanced or recurrent head and neck cancer (HNC) .

* To determine the recommended light irradiance dose for a future Phase 2 trial of Photofrin® mediated I-PDT in patients with locally advanced or recurrent HNC

EXPLORATORY OBJECTIVES:

I . To access the objective tumor response rate

OUTLINE: This is a phase I study .

Patients receive porfimer sodium intravenously (IV) over 3-5 minutes and undergo I-PDT approximately 48 hours later.

After completion of study treatment, patients are followed up every 1-3 months for the first year, 2-6 months for 2nd year, and annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Patients with locally advanced or recurrent head and neck cancer who failed to respond to standard therapy and are not amenable to standard curative treatment.
* Tumor accessible for unrestricted illumination for interstitial photodynamic therapy (PDT) (accessibility as determined by the physician).
* Life expectancy of at least 6 months, in the judgment of the physician.
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Subject must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* High dose curative radiotherapy within 30 days in the area to be treated. Tumor invading a major blood vessel.
* Tumor is not measurable on a computed tomography (CT) or magnetic resonance imaging (MRI) scan according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Location and extension of the tumor precludes a potentially effective I-PDT.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with porphyria, or with known hypersensitivity to porphyrins or porphyrin-like compounds.
* Platelet count < 75,000.
* Total serum bilirubin > 2 mg/dL
* Alkaline phosphatase (hepatic) > 3 times the upper normal limit
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 3 times the upper normal limit
* Patients with moderately to severely impaired creatinine clearance (crcl < 44) will be excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female subjects.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive porfimer sodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Wooten, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A(Porfimer Sodium, I-PDT
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Arm A(Porfimer Sodium, I-PDT
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: The frequency of toxicities will be tabulated by max grade of any Adverse Events experience by a patient across dose levels and cycles. All subjects who receive any study treatment will be considered evaluable for toxicity.
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A(Porfimer Sodium, I-PDT
Number analyzed (Participants) | 5
Participants
  grade 1 | 0
  grade 2 | 1
  grade 3 | 4
  grade 4 | 0

ADVERSE EVENTS:
Time Frame: Routine visits at 10-12 weeks and until 8 months
Arm/Group | Arm A(Porfimer Sodium, I-PDT
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A(Porfimer Sodium, I-PDT (N=5)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Social circumstances - Other, specify (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A(Porfimer Sodium, I-PDT (N=5)
Photophobia (Eye disorders) | 1 (1)
Vision decreased (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (3)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT03727061/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT03727061/ICF_000.pdf